CLINICAL TRIAL: NCT03507244
Title: Intrathecal-pemetrexed Combined With Concurrent Involved-field Radiotherapy for Leptomeningeal Metastasis From Solid Tumor: a Phase I/II Clinical Trial
Brief Title: Concurrent Intrathecal-pemetrexed and Involved-field Radiotherapy for Leptomeningeal Metastasis From Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Zhenyu Pan, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPLM
Record Dates: First submitted 2018-03-31; First posted 2018-04-25 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Leptomeningeal Metastasis
Keywords: Leptomeningeal metastasis; Malignant solid tumors; Pemetrexed; Intrathecal chemotherapy; Radiotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis | interventions — Pemetrexed; Dexamethasone; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group 1,Intra-pemetrexed, radiotherapy (Experimental): The treatment regimen consisted of intrathecal chemotherapy (via lumbar puncture, pemetrexed 10 mg, plus dexamethasone 5 mg, once per week, 5-8 times, 4-7 weeks in total) and radiotherapy. Radiotherapy consisted of fractionated, conformal radiation given at a daily dose of 2 Gy. The planning volume consisted of sites of symptomatic disease, bulky disease observed on magnetic resonance imaging, including the whole brain and basis cranii received 40 Gy in 20 fractions, 4 weeks in total, and/or segment of spinal canal received 40-50 Gy.
  Interventions: Drug: Pemetrexed; Drug: Dexamethasone; Radiation: Radiotherapy

INTERVENTIONS:
Drug: Pemetrexed — Pemetrexed, 10 mg,intrathecal injection, plus dexamethasone 5 mg, once per week, 5 to 8 times, 4 to 7 weeks in total.
Drug: Dexamethasone — Dexamethasone, 5 mg, intrathecal injection, simultaneously with pemetrexed, once per week, 5 to 8 times, 4 to 7 weeks in total.
Radiation: Radiotherapy — The sites of symptomatic disease, bulky disease observed on MRI, including the whole brain and basis cranii, 40 Gy in 20 fractions;and/or segment of spinal canal received 40-50 Gy in 20-25 fractions.

SUMMARY:
Intrathecal chemotherapy is one of the most important treatment modalities for leptomeningeal metastasis of solid tumors. In the previous retrospective study, it has been proved that concurrent radiotherapy and intrathecal methotrexate for leptomeningeal metastasis from solid tumors with adverse prognostic factors showed great effectiveness and safety. The preliminary results of investigators' current prospective clinical study (Involved-field Radiotherapy Combined With Concurrent Intrathecal-methotrexate Versus Intrathecal-Ara-C for Leptomeningeal Metastases From Solid Tumor: A Randomized Phase II Clinical Trial. ClinicalTrials.gov identification number: NCT03082144) also showed that the regimen of concurrent intrathecal chemotherapy and radiotherapy may serve as an optimal therapeutic option for treatment of leptomeningeal metastases from solid tumors. Pemetrexed is a newer multitargeted antifolate which has shown activity in various tumors. In investigators' current study (Intrathecal Pemetrexed for Recurrent Leptomeningeal Metastasis From Non-small Cell Lung Cancer: A Prospective Pilot Clinical Trial. ClinicalTrials.gov identification number: NCT03101579), the regimen of intrathecal pemetrexed with folic acid and vitamin B12 supplementation may provide higher effectiveness and safety for recurrent leptomeningeal metastasis from non-small cell lung cancer. Therefore, the purpose of the study is to evaluate the tolerability, safety and effectiveness of intrathecal pemetrexed combined with involved-field radiotherapy as the first line treatment in patients with leptomeningeal metastases from malignant solid tumors.

DETAILED DESCRIPTION:
This study is a single arm, open clinical trial. Consecutive patients with leptomeningeal metastases from malignant solid tumors are enrolled into this study. Concomitant regimen consisted of intrathecal chemotherapy (via lumbar puncture, pemetrexed 10 mg, plus dexamethasone 5 mg, once per week, 5 to 8 times, 4 to 7 weeks in total) and radiotherapy. Radiotherapy consisted of fractionated, conformal radiation given at a daily dose of 2 Gy. The planning volume consisted of sites of symptomatic disease, bulky disease observed on magnetic resonance imaging(MRI), including the whole brain and basis cranii received 40 Gy in 20 fractions, 4 weeks in total, and/or segment of spinal canal received 40-50 Gy. The RANO proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have been definitely diagnosed as leptomeningeal metastasis according to cerebrospinal fluid (CSF) cytology, or patients who got the clinical diagnosis by combining history of cancer, neuroimaging, clinical manifestation, and CSF examination, etc.
2. Patients who have been diagnosed as malignant solid tumor with definite pathologic type, excluding hematological malignancies (e.g., leukemia and lymphoma) or intracranial germ cell tumors;
3. No severe abnormal liver function; normal kidney function; WBC≥4000/mm3, Plt≥110000/mm3;
4. No other severe chronic diseases;
5. No severe dyscrasia.

Exclusion Criteria:

1. Patients with leptomeningeal metastasis from unknown primary tumor;
2. Patients who had received whole brain radiotherapy in the past 10 months;
3. Patients who had accepted systemic chemotherapy within two weeks, or molecular targeted therapy less than two weeks;
4. Patients with poor compliance, or for other reasons, the researchers considered unsuitable to participate in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-01-15 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events | The evaluation was performed at 3 months after the end of treatment or when patient died.
  The incidence of treatment-related adverse events were measured for determing tolerability and safety. Adverse events (AEs) are evaluated according to the Common Terminology Criteria for Adverse Events (CTCAE, version 4.03). Events of grade 3-5 are defined as moderate and severe adverse events.

SECONDARY OUTCOMES:
Clinical response rate | The evaluation was performed at 3 months after the end of treatment or when patient died.
  The RANO proposal for response criteria of leptomeningeal metastasis was used to assess the clinical response in this study.
Overall survival | The evaluation was performed at least 7 months after leptomeningeal metastasis diagnosis or until death.
  Survival time was recorded since the date of patient enrollment. All patients were followed up until death or the end of the study.
Neurological progression-free survival (NPFS) | All patients were followed up at least 6 months, and the evaluation of NPFS was performed from the beginning of treatment until the date of first documented neurological progression or date of death from any cause, whichever came first.
  NPFS was defined as time from the start of treatment until neurological progression or death. The neurological progression was determined based on the RANO proposal evaluation criteria which have been established and published on Neuro Oncol.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Pan, Professor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

REFERENCES:
- [Result] Pan Z, Yang G, He H, Zhao G, Yuan T, Li Y, Shi W, Gao P, Dong L, Li Y. Concurrent radiotherapy and intrathecal methotrexate for treating leptomeningeal metastasis from solid tumors with adverse prognostic factors: A prospective and single-arm study. Int J Cancer. 2016 Oct 15;139(8):1864-72. doi: 10.1002/ijc.30214. Epub 2016 Jun 30. PMID 27243238
- [Result] Stoop MP, Visser S, van Dijk E, Aerts JGJV, Stricker BH, Luider TM. A new quantification method for assessing plasma concentrations of pemetrexed and its polyglutamate metabolites. J Pharm Biomed Anal. 2016 Sep 5;128:1-8. doi: 10.1016/j.jpba.2016.04.036. Epub 2016 Apr 30. PMID 27209449
- [Result] Chattopadhyay S, Moran RG, Goldman ID. Pemetrexed: biochemical and cellular pharmacology, mechanisms, and clinical applications. Mol Cancer Ther. 2007 Feb;6(2):404-17. doi: 10.1158/1535-7163.MCT-06-0343. PMID 17308042
- [Result] Sorensen JB. Pharmacokinetic evaluation of pemetrexed. Expert Opin Drug Metab Toxicol. 2011 Jul;7(7):919-28. doi: 10.1517/17425255.2011.587411. Epub 2011 May 21. PMID 21599552
- [Result] Adjei AA. Pharmacology and mechanism of action of pemetrexed. Clin Lung Cancer. 2004 Apr;5 Suppl 2:S51-5. doi: 10.3816/clc.2004.s.003. PMID 15117425
- [Result] Mita AC, Sweeney CJ, Baker SD, Goetz A, Hammond LA, Patnaik A, Tolcher AW, Villalona-Calero M, Sandler A, Chaudhuri T, Molpus K, Latz JE, Simms L, Chaudhary AK, Johnson RD, Rowinsky EK, Takimoto CH. Phase I and pharmacokinetic study of pemetrexed administered every 3 weeks to advanced cancer patients with normal and impaired renal function. J Clin Oncol. 2006 Feb 1;24(4):552-62. doi: 10.1200/JCO.2004.00.9720. Epub 2006 Jan 3. PMID 16391300
- [Result] McDonald AC, Vasey PA, Adams L, Walling J, Woodworth JR, Abrahams T, McCarthy S, Bailey NP, Siddiqui N, Lind MJ, Calvert AH, Twelves CJ, Cassidy J, Kaye SB. A phase I and pharmacokinetic study of LY231514, the multitargeted antifolate. Clin Cancer Res. 1998 Mar;4(3):605-10. PMID 9533527
- [Result] Rinaldi DA, Kuhn JG, Burris HA, Dorr FA, Rodriguez G, Eckhardt SG, Jones S, Woodworth JR, Baker S, Langley C, Mascorro D, Abrahams T, Von Hoff DD. A phase I evaluation of multitargeted antifolate (MTA, LY231514), administered every 21 days, utilizing the modified continual reassessment method for dose escalation. Cancer Chemother Pharmacol. 1999;44(5):372-80. doi: 10.1007/s002800050992. PMID 10501910
- [Result] Stapleton SL, Reid JM, Thompson PA, Ames MM, McGovern RM, McGuffey L, Nuchtern J, Dauser R, Blaney SM. Plasma and cerebrospinal fluid pharmacokinetics of pemetrexed after intravenous administration in non-human primates. Cancer Chemother Pharmacol. 2007 Mar;59(4):461-6. doi: 10.1007/s00280-006-0285-7. Epub 2006 Jul 20. PMID 16855840
- [Result] Kumthekar P, Grimm SA, Avram MJ, Kaklamani V, Helenowski I, Rademaker A, Cianfrocca M, Gradishar W, Patel J, Mulcahy M, McCarthy K, Raizer JJ. Pharmacokinetics and efficacy of pemetrexed in patients with brain or leptomeningeal metastases. J Neurooncol. 2013 Apr;112(2):247-55. doi: 10.1007/s11060-013-1055-0. Epub 2013 Jan 25. PMID 23354655
- [Derived] Pan Z, Yang G, He H, Cui J, Li W, Yuan T, Chen K, Jiang T, Gao P, Sun Y, Cong X, Li Z, Wang Y, Pang X, Song Y, Zhao G. Intrathecal pemetrexed combined with involved-field radiotherapy as a first-line intra-CSF therapy for leptomeningeal metastases from solid tumors: a phase I/II study. Ther Adv Med Oncol. 2020 Jul 17;12:1758835920937953. doi: 10.1177/1758835920937953. eCollection 2020. PMID 32733606